CLINICAL TRIAL: NCT00666510
Title: Higher Exhaled Nitric Oxide (NO) is Associated With Intraoperative Bronchospasm
Brief Title: Bronchospasm Associated With High Nitric Oxide
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Joaquim Edson Vieira, Fisiopatologia Experimental FMUSP
Other Study IDs: CAP125-01
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Asthma; Airway Hyperresponsiveness
Keywords: nitric oxide; bronchospasm; anesthesia; induced sputum; asthma
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity; Bronchial Spasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bronchospasm: Patients who presented bronchospasm during anesthesia induction
- Asthma: Patients who presented bronchospasm during anesthesia induction and were identified as asthmatics
- Control: Patients who were submitted to anesthesia induction and showed no complications

SUMMARY:
Intraoperative bronchospasm challenges anesthesia's safety. This study aims to investigate high concentration of exhaled nitric oxide as a marker of intraoperative bronchospasm.

DETAILED DESCRIPTION:
Previous studies in asthmatic patients suggested that exhaled nitric oxide may represent a noninvasive measure for airway inflammation. Anesthesia information forms from 1999 throughout 2004 were revised (n=146.358). Bronchospasm occurrence appeared registered on 863 forms. From those, nine were identified as non-asthmatics patients (Bronchospasm group). Also, 12 asthmatics constituted one additional group (Asthma group) and 10 subjects with no previous airway disease or symptoms (Control group). All subjects were submitted to Exhaled nitric oxide measurements (parts/billion), spirometry and induced sputum.

ELIGIBILITY:
Inclusion Criteria:

* patients with no systemic disease and registered bronchospasm during anesthesia induction

Exclusion Criteria:

* hypertension, COPD, diabetes, pregnancy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital, late post-anesthesia cared patients
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 1999-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide in parts per billion | one to six months after surgery

SECONDARY OUTCOMES:
Eosinophils concentration within sputum sample, pulmonary function tests | one to six months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, MD, PhD, Principal Investigator — University of Sao Paulo Medical School - FMUSP
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil